CLINICAL TRIAL: NCT04677647
Title: OurChild: A Health IT Solution to Reduce Minority Health Disparities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-01468
Record Dates: First submitted 2020-12-17; First posted 2020-12-21 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Mental Health
Keywords: Health Information Technology
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OurChild (Experimental)
  Interventions: Other: OurChild mHealth Digital Platform

INTERVENTIONS:
Other: OurChild mHealth Digital Platform — The intervention being created and tested in this study is OurChild an integrated mHealth/EHR app, initially designed for the Chinese American community in Sunset Park, Brooklyn. All participants will be assigned to either beta versions undergoing development, or to version 1.0.

SUMMARY:
Chinese American immigrant families are a fast-growing immigrant group with unmet early childhood mental health needs. The team proposes to design, build, and implement OurChild, an integrated mHealth/EHR solution to increase access to early childhood mental health knowledge and mental health services and resources for Chinese American children ages 2-6 years old and their parents in the Sunset Park Brooklyn.

DETAILED DESCRIPTION:
The goal of this study is to reduce health disparities by designing a digital solution (OurChild) that facilitates connection and bidirectional exchange of information across the cultural, contextual, language, and setting differences that are key barriers to early childhood mental health knowledge and care access for the Chinese American community in Sunset Park, Brooklyn. The first study aim is to iteratively design, build, and test OurChild. To do this, the team will 1) collaborate with family, clinical, and community stakeholders to conduct an early childhood mental health context/needs analysis and participatory design and discovery activities; 2) build a digital library of early childhood mental health resources accessible from OurChild; and 3) pilot and assess the usability and acceptability of a beta version of OurChild in a mixed-methods, cross-sectional cohort of 12 Chinese American parents and their 2- to 6-year-old children (N=24) who receive care at the Sunset Park 7th Avenue Family Health Center; and 5) optimize the design, features, and performance to create OurChild 1.0. The second study aim is to evaluate the reach, effectiveness, adoption, implementation and maintenance of OurChild 1.0 through an implementation cohort study with 120 parent/child dyads (N=240). A mixed-methods approach using metadata collected with the OurChild app, parent-reported data from the app, EHR data, and post-implementation key informant interviews with providers and other stakeholders to determine whether use of OurChild increases referrals of young children for a mental health consultation or evaluation (Primary Aim) will be used. The secondary aims include examining whether use of OurChild increases 1) parent self-efficacy; 2) parent-provider engagement; and 3) linkage with community early childhood resources.

ELIGIBILITY:
Inclusion Criteria:

* Child must be 24 to 72 months old
* Child must have been receiving pediatric primary care at the 7th Ave FHC for at least 6 months
* Child must be identified as Chinese and/or preferred language is Chinese in EHR
* Parents must be at least 18 years old
* Parents must be the child's parent/legal guardian
* Parents must be able and willing to provide informed consent

Exclusion Criteria:

* Siblings and parents of previously enrolled children
* Parents who do not have access to an iOS or Android smartphone

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2023-07-25 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Number of Referrals | Month 18, Month 45
  Change in number of referrals to NYU Langone Child Psychiatry or Developmental Pediatrics

SECONDARY OUTCOMES:
Change in Score on Parental Self-Efficacy Scale | Month 25, Month 45
  The General Self-Efficacy Scale is a 10-item psychometric scale that is designed to assess optimistic self-beliefs to cope with a variety of difficult demands in life.
Change in Amount of parent-provider engagement | Month 18, Month 45
  Engagement defined as at least one interaction or messaging exchange between parent and provider through OurChild messaging portal
Change in accessing resources on App | Month 25, Month 45
  Access to clinical and community early childhood and family services and resources; access defined as click through on resources library tab in OurChild app
Score on Betz Physician Confidence Scale | Month 48
  The Betz Scale is a collection of 11 statements describing the provider's perceived barriers to the identification and management of child mental health issues. Responses to each statement consist of Strongly Agree (0), Agree, Uncertain, Disagree, and Strongly Disagree (5). The total range of score is 0-55, with a higher score indicating higher physician confidence in assessing and treating mental health disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Simona Kwon, DrPH, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to helen.egger@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.